CLINICAL TRIAL: NCT05124769
Title: Allowing Pain Versus Avoiding Pain During Shoulder Exercises: Does Pain Matter in the Effectiveness of an Exercise Program in Patients With Rotator Cuff Tendinopathy?
Brief Title: PAin During Shoulder Exercise
Acronym: PASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Birgitte Hougs Kjær, Principal investigator, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BispebjergH_PASE_BKjaer
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-12

CONDITIONS: Rotator Cuff Tendinopathy
Keywords: rotator cuff; tendinopathy; tendinosis; shoulder; overuse injuries
MeSH Terms: conditions — Tendinopathy; Cumulative Trauma Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with parallel assignment
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double (investigator, outcome assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Allow (Experimental): Pain is allowed up to 5/10 during exercises, monitored by NPRS. Depending on tissue irritability and other factors such as ROM, the exercises may be performed in an isometric way, or dynamic.
  Interventions: Behavioral: Pain Allowing Program (PAllow)
- Pain Avoid (Active Comparator): Pain is not allowed during the exercises, and should be <2/10, monitored by NPRS.
  Interventions: Behavioral: Pain Avoiding Program (PAvoid)

INTERVENTIONS:
Behavioral: Pain Allowing Program (PAllow) — Performing exercises considered to have a considerable supraspinatus/ infraspinatus tendon/muscle load (EMG muscle activity of > 40% MVC).
  Arms: Pain Allow
Behavioral: Pain Avoiding Program (PAvoid) — Performing exercises selected to have a minimal insupraspinatus/ infraspinatus tendon/muscle load (EMG muscle activity of <20% MVC).
  These unloading exercises are performed for 6 weeks. In the second part of the exercise protocol, the "loading" exercises are applied, however without pain.
  In case the patient still feels pain during the exercises in that period, the "unloading" exercises are continued.
  Arms: Pain Avoid

SUMMARY:
Overuse shoulder injuries such as rotator cuff (RC) tendinopathy are common with a prevalence estimated to be 14% in the general population of which 23% of the working population with shoulder problems are sick listed.

RC tendinopathy is a tendon-related pain in the proximal lateral aspect of the upper arm with weakness, especially during active elevation and external rotation, and painful active range of motion. The prevalence of RC tendinopathy is highest in the supraspinatus and infraspinatus tendon.

Exercise therapy is regarded as an effective intervention for symptomatic RC tendinopathy for reducing pain and disability and improving function. However, the prescription is diverse and the effectiveness of specific characteristics of exercise programs is unknown. Many contextual factors and prescription parameters, such as external resistance, training intensity and frequency, home versus supervised exercises, duration of the program, etc. have been described. Some of these prescription parameters have been extensively studied, with some conflicting results. Although some level of resistance seems to matter, as well as number of sets and repetitions, the 'optimal' level and volume are unclear. Inducing or allowing pain based on tendon loading during exercises is todays consensus in the treatment of patellar and achilles tendinopathy using a pain-monitoring model. Although a number of shoulder studies report that pain either should be avoided or allowed, not one study ever examined the influence of pain allowance versus pain avoidance during a shoulder exercise program on patient outcome in terms of pain, physical function and disability.

The purpose of this project is to examine the effect of allowing pain versus avoiding pain based on tendon loading during an exercise regimen for patients with symptomatic rotator cuff (RC) tendinopathy. This will be accomplished in a Randomized Controlled Clinical Trial, comparing the effectiveness on patient reported and objective outcomes of a "pain allowing" and "pain avoiding" exercise program, performed for 26 weeks. Our hypothesis is that allowing pain based on tendon loading during exercises would result in a better outcome in pain and function measured on SPADI (the primary outcome) compared to avoiding pain in patients with RC tendinopathy.

DETAILED DESCRIPTION:
Aim The purpose of this project is to examine the effect of allowing pain versus avoiding pain based on tendon loading during an exercise regimen for patients with symptomatic rotator cuff (RC) tendinopathy. This will be accomplished in a Randomized Controlled Clinical Trial, comparing the effectiveness on patient reported and objective outcomes of a "pain allowing" and "pain avoiding" exercise program, performed for 26 weeks.

Background Shoulder disorders are the third most common musculoskeletal disorder with a life-time prevalence in the general population of 30%. Shoulder disorders are often persistent and recurrent, with 54% of the patients reporting on-going symptoms after 3 years. RC tendinopathy is regarded as a common source of shoulder pain with prevalence estimated to be as high as 14% in the general working-age population. About 23% of the working population with shoulder problems are sick-listed, with a potential individual productivity loss.

RC tendinopathy is a tendon-related pain in the proximal lateral aspect of the upper arm with weakness, especially during active elevation and external rotation, and painful active range of motion. The pathoanatomic understanding is extended by classifying tissue irritability and specific impairments. Tissue irritability is meant to guide intensity of treatment, and identifying specific impairments guides specific tactics used for intervention. The prevalence of RC tendinopathy is highest in the supraspinatus and infraspinatus tendon.

Exercise therapy is widely regarded as an effective intervention for symptomatic RC tendinopathy for reducing pain and disability and improving function. It is well known that tendon collagen regains formation and tensile strength faster than unstressed collagen, and that it can take 12 month or longer before it reaches full maturity and strength. However, the prescription is diverse and the effectiveness of specific characteristics of exercise programs is unknown. Many contextual factors and prescription parameters, such as external resistance, training intensity and frequency, home versus supervised exercises, duration of the program, etc. have been described and are summarized in a systematic review. Some of these prescription parameters have been extensively studied, with some conflicting results. Although some level of resistance seems to matter, as well as a number of sets and repetitions, the 'optimal' level and volume are unclear. The existing studies offer some preliminary guidance in relation to the development and application of loading in exercise programs for RC tendinopathy, however there is a gap in literature with respect to allowing or avoiding pain during shoulder exercises. Inducing or allowing pain based on tendon loading during exercises is todays consensus in the treatment of patellar and achilles tendinopathy using a pain-monitoring model.

Although a number of shoulder studies report that pain either should be avoided or allowed, not one study ever examined the influence of pain allowance versus pain avoidance during a shoulder exercise program on patient outcome in terms of pain, physical function and disability.

Hypothesis Allowing pain based on tendon loading during exercises would result in a better outcome in pain and function measured on SPADI (the primary outcome) compared to avoiding pain in patients with RC tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 55 years
* Shoulder symptoms lasting for a minimum of 3 months
* Clinical diagnosis of rotator cuff (supraspinatus and/or infraspinatus) tendinopathy
* Clinical diagnosis verified by/ combined with ultrasound

Exclusion Criteria:

Patients are excluded if they have

* resting pain above 4/10 (NPRS)
* <90 degrees active elevation of the arm
* had a corticosteroid injection within the previous 12 weeks
* isolated subscapularis tendinopathy
* total rotator cuff tear
* diagnosed AC-joint pathology
* diagnosed labrum pathology
* diagnosed glenohumeral joint instability
* had prior shoulder surgery (all shoulder joints)
* diagnosed glenohumeral osteo arthrosis (OA) evaluated on x-ray, rheumatoid arthritis or periarthrosis General exclusion criteria are inability to speak or read Danish, inability to perform and maintain the physical training, or other conditions negatively influencing compliance.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Shoulder Pain and Disability Index (SPADI) | 26-week
  Self-reported measure of pain and function. The responses are indicated on a visual analogue scale where 0 = no pain/no difficulty and 10 = worst imaginable pain/so difficult it requires help. The items are summed and converted to a total score out of 100 where a high score indicates greater pain and disability in patients with shoulder disorders.

SECONDARY OUTCOMES:
Change from baseline in Shoulder Pain and Disability Index (SPADI) | 52-week
  Self-reported measure of pain and function. The responses are indicated on a visual analogue scale where 0 = no pain/no difficulty and 10 = worst imaginable pain/so difficult it requires help. The items are summed and converted to a total score out of 100 where a high score indicates greater pain and disability in patients with shoulder disorders.
Change from baseline in Disabilities Arm, Shoulder and Hand questionnaire (DASH) | 26 and 52 weeks
  Self-reported measure of pain, function and quality of life. The questionnaire score ranges from 0 to 100 where 0 equals no disability and 100 equals the most severe disability.
Change from baseline in Numeric Pain Rating Scale (NPRS) | 26 and 52 weeks
  Self-reported measure of pain. The score ranges from 0 to 10 where 0 equals no pain and 10 equals the most severe pain.
Patient Acceptable Symptom State (PASS) | 6, 26 and 52 weeks
  Self-reported measure of symptom acceptability. The PASS threshold is determined by asking patients if they are satisfied with their current health state. Patients respond to this question with "yes" or "no".
Global Rating Scale (GRS) | 6, 26 and 52 weeks
  Self-reported measure of change of condition. The GRS is used to obtain a general impression of recovery from baseline to 26 and 52 weeks after baseline with the question: "Compared to when this treatment first started, how would you describe your shoulder this last week?" This is assessed on a 15-point scale where - 7 represents vastly worse, 0 represents unchanged, and + 7 represents much better.
Change from baseline in Range-of-motion (ROM) in scapular plane elevation (standing) and in external (supine in 90° abduction) | 26 and 52 weeks
  Objective measure
Change from baseline in Isometric muscle strength (MVC) in shoulder elevation in scapular plane and external shoulder rotation | 26 and 52 weeks
  Objective measure

OTHER OUTCOMES:
Change from baseline in Pressure Pain Threshold (PPT) | 26 weeks
  Objective measure
Quantitative and qualitative ultrasound (US) evaluation | Baseline, 26 and 52 weeks
  Objective measure
Workability Index (WAI) | Baseline, 26 and 52 weeks
  Working ability A single item question concerning current work ability compared with the lifetime best, with a possible score 0 ('completely unable to work') to 10 ('work ability at its best').
Sport participation | Baseline, 26 and 52 weeks
  Sport participation and return to sport

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte H Kjær, Ph.D, Principal Investigator — Bispebjerg and Frederiksberg Hospitals
Locations (1):
- Bispebjerg and Frederiksberg Hospital, Copenhagen NV, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kjaer BH, Cools AM, Johannsen FE, Trostrup J, Bieler T, Siersma V, Magnusson PS. To allow or avoid pain during shoulder rehabilitation exercises for patients with chronic rotator cuff tendinopathy-Study protocol for a randomized controlled trial (the PASE trial). Trials. 2024 Feb 21;25(1):135. doi: 10.1186/s13063-024-07973-6. PMID 38383459

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-12-19): https://cdn.clinicaltrials.gov/large-docs/69/NCT05124769/SAP_001.pdf